CLINICAL TRIAL: NCT05581134
Title: Effectiveness of Immersive Virtual Reality Rehabilitation Program to Reduce Symptoms Severity and Improve Quality of Life in Patients With Functional Motor Disorders
Brief Title: Immersive Virtual Reality in Functional Motor Disorders
Acronym: FMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marialuisa Gandolfi (Other)
Responsible Party: Sponsor-Investigator, Marialuisa Gandolfi, MD, PhD, Universita di Verona
Organization: Universita di Verona (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JP-VR-19
Record Dates: First submitted 2022-10-01; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Functional Motor Disorders
Keywords: Virtual Reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: An examiner blinded to group allocation will assess all patients. To keep blindness, the examiner will not ask for information about the treatment to the patients or the caregivers, and this last will be instructed not to give any extra information outside of the examiner's questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Patients will attend the in-person 5-day rehabilitation program (2 h/day) to re-establish normal movement patterns in a dynamic and challenging VR environment. During each session, the patients will be supervised by the physiotherapist. The immersive VR system will simultaneously deliver visual and auditory distractors during the exercises.
  Interventions: Device: Virtual Reality intervention
- Control Group Treatment (Active Comparator): Patients will attend the in-person 5-day rehabilitation program (2 h/day) to re-establish normal movement patterns within a multidisciplinary etiological framework according to a validated rehabilitation protocol for FMDs.The conventional group will undergo the same dose, frequency, and intensity of rehabilitation treatment as the VR group consisting of rehabilitation without VR exercises.
  Interventions: Behavioral: Control Group intervention

INTERVENTIONS:
Device: Virtual Reality intervention — Virtual reality (VR) is a powerful tool to create an illusory state in which the user can feel that they have been transported to a new location (place illusion), that events happening are real (plausibility illusion), and even that bodies have been substituted by an avatar (embodiment illusion). VR illusions are driven by the same neurological mechanisms of everyday perception of the body in the world and induce realistic responses to VR.
  Arms: Virtual Reality Group
Behavioral: Control Group intervention — Treatment will follow general treatment principles in physiotherapy for FMDs: (1) education; (2) exploration of how symptoms affect movement and posture; (3) retraining movement using strategies based on redirection of attention; and (4) development of a self-management plan.
  Arms: Control Group Treatment

SUMMARY:
The study aims to demonstrate the effectiveness and superiority of a 5-day immersive VR-rehabilitation treatment versus a 5-day conventional rehabilitation treatment in reducing FMDs symptoms severity, assessed by the Simplified Functional Movement Disorders Rating Scale (S- FMDRS).

DETAILED DESCRIPTION:
This is a single-blind, randomized controlled trial to evaluate the superiority of immersive VR distractors combined with graded physical exercises over conventional rehabilitation (without any VR distractors) to reduce FMDs symptoms and improve gait and balance. Patients will be randomized to receive the experimental training (VRG) or the control training (CRG) (allocation ratio 1:1). The primary and secondary outcomes will be measured by the same examiner before (T0), at the end of the treatment (T1), and at three-month follow-up after the end of the treatment (T2). The test order will be the same across all evaluation sessions. The examiner will be blinded to group assignments.

ELIGIBILITY:
Inclusion criteria were: established diagnosis of FMDs, age ≥ 18 years, and acceptance of the diagnosis.

Exclusion criteria were: prominent dissociative seizures, prominent cognitive and/or physical impairment that precluded signing the informed consent form for study participation based on clinical judgment, incomplete assessment, and questionnaire because of language comprehension difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-29 (Estimated)

PRIMARY OUTCOMES:
Change in the Simplified Functional Movement Disorders Rating Scale (S-FMDRS) score | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  Objective-rated validated scale to rate the duration and severity of functional motor symptoms (range: 0-54; higher = worse).

SECONDARY OUTCOMES:
Change in the Multidimensional Fatigue Inventory Scale (MFI-20) score | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  It evaluates fatigue differentiating general, physical, reduced-activity, reduced-motivation, and mental fatigue (subscale range: 4-20; higher = worse).
Change in the Brief Pain Inventory (BPI) score | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  It evaluates pain intensity (range: 0-40; higher = worse) and interference (range: 0-70; higher = worse).
Change in the Beck Depression Inventory (BDI-II) score | Before the intensive 5-day rehabilitation program (T0) and after 12 weeks (T2).
  It evaluates depression (range: 0-63; higher = worse).
Change in the Beck Anxiety Inventory (BAI) score | Before the intensive 5-day rehabilitation program (T0) and after 12 weeks (T2).
  It evaluates anxiety (range: 0-63; higher = worse).
Change in the 12-item Short-Form Health Survey (SF-12) score | Before the intensive 5-day rehabilitation program (T0) and after 12 weeks (T2).
  The health-Related QoL will be evaluated by the Mental Health and Physical functioning of the 12-item Short-Form Health Survey (SF-12) (range: 0-100; higher = better)
Change in the Clinical Global Impression (CGI) score | Before the intensive 5-day rehabilitation program (T0) and after 12 weeks (T2).
  Self-rated perception of change will be assessed with the 7-point Clinical Global Impression (CGI) scale with scores from 1 (very much improved) to 7 (very much worse).
Change in gait speed (cm/sec) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  Gait analysis will be used to collect gait speed (cm/s).
Change in Swing time (%) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  Gait analysis will be used to collect swing time (%).
Change in Stride time (s) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  Gait analysis will be used to collect stride time (s).
Change in Stride length (cm) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  Gait analysis will be used to collect stride length (cm).
Change in sway area (mm2) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  An electronic monaxial stabilometric platform will be used to collect sway area (mm2).
Change in total excursion path (mm) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  An electronic monaxial stabilometric platform will be used to collect total excursion path (mm).
Change in velocity of Cop displacement in the anteroposterior directions (mm/s) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  An electronic monaxial stabilometric platform will be used to collect the velocity of Cop displacement in the anteroposterior directions.
Change in velocity of Cop displacement in the mediolateral directions (mm/s) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1), and after 12 weeks (T2).
  An electronic monaxial stabilometric platform will be used to collect the velocity of Cop displacement in the mediolateral directions.
Change in the Toronto Alexithymia Scale (TAS-20) score | Before the intensive 5-day rehabilitation program (T0) and after 12 weeks (T2).
  It evaluates the level of alexithymia (range: 20-100; higher = worse)

OTHER OUTCOMES:
Number of drop-out | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1)
  The number of dropouts before the end of treatment will be collected. The experimental group will report adverse events on the use of VR.
number of patients who refuse the treatment | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1)
  Recruitment rate
number of falls or event near falling | after the intensive 5-day rehabilitation program (T1)
  Falls or event near falling occurred during the rehabilitation in both groups
Score on the Simulation Sickness Questionnaire (SSQ) | Before the intensive 5-day rehabilitation program (T0), after the intensive 5-day rehabilitation program (T1)
  It will be used to evaluate the level of symptoms associated with simulator sickness (subscale range: 0-48; higher=worse)

CONTACTS AND LOCATIONS:
Overall Officials: Marialuisa Gandolfi, PhD, Principal Investigator — Università di Verona
Locations (1):
- Department of Neurosciences, Biomedicine and Movement Sciences, University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nielsen G, Buszewicz M, Stevenson F, Hunter R, Holt K, Dudziec M, Ricciardi L, Marsden J, Joyce E, Edwards MJ. Randomised feasibility study of physiotherapy for patients with functional motor symptoms. J Neurol Neurosurg Psychiatry. 2017 Jun;88(6):484-490. doi: 10.1136/jnnp-2016-314408. Epub 2016 Sep 30. PMID 27694498
- [Background] Lubetzky AV, Kary EE, Harel D, Hujsak B, Perlin K. Feasibility and reliability of a virtual reality oculus platform to measure sensory integration for postural control in young adults. Physiother Theory Pract. 2018 Dec;34(12):935-950. doi: 10.1080/09593985.2018.1431344. Epub 2018 Jan 24. PMID 29364733
- [Background] Kim A, Darakjian N, Finley JM. Walking in fully immersive virtual environments: an evaluation of potential adverse effects in older adults and individuals with Parkinson's disease. J Neuroeng Rehabil. 2017 Feb 21;14(1):16. doi: 10.1186/s12984-017-0225-2. PMID 28222783
- [Background] Nielsen G, Stone J, Matthews A, Brown M, Sparkes C, Farmer R, Masterton L, Duncan L, Winters A, Daniell L, Lumsden C, Carson A, David AS, Edwards M. Physiotherapy for functional motor disorders: a consensus recommendation. J Neurol Neurosurg Psychiatry. 2015 Oct;86(10):1113-9. doi: 10.1136/jnnp-2014-309255. Epub 2014 Nov 28. PMID 25433033
- [Background] Perez DL, Edwards MJ, Nielsen G, Kozlowska K, Hallett M, LaFrance WC Jr. Decade of progress in motor functional neurological disorder: continuing the momentum. J Neurol Neurosurg Psychiatry. 2021 Mar 15:jnnp-2020-323953. doi: 10.1136/jnnp-2020-323953. Online ahead of print. PMID 33722822
- [Result] Gandolfi M, Sandri A, Geroin C, Bombieri F, Riello M, Menaspa Z, Bonetto C, Smania N, Tinazzi M. Improvement in motor symptoms, physical fatigue, and self-rated change perception in functional motor disorders: a prospective cohort study of a 12-week telemedicine program. J Neurol. 2022 Nov;269(11):5940-5953. doi: 10.1007/s00415-022-11230-8. Epub 2022 Jul 9. PMID 35809125
- [Result] Gandolfi M, Riello M, Bellamoli V, Bombieri F, Geroin C, Di Vico IA, Tinazzi M. Motor and non-motor outcomes after a rehabilitation program for patients with Functional Motor Disorders: A prospective, observational cohort study. NeuroRehabilitation. 2021;48(3):305-314. doi: 10.3233/NRE-201617. PMID 33780378